CLINICAL TRIAL: NCT01395797
Title: Effects of Pioglitazone, a PPARγ Agonist, on the Abuse Liability of Heroin and of Nicotine
Brief Title: Pioglitazone for Heroin and for Nicotine Dependence
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The funding period ended.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 6255; R01DA031022 (NIH)
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Heroin Dependence; Nicotine Dependence
MeSH Terms: conditions — Heroin Dependence; Tobacco Use Disorder | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo - Heroin (Placebo Comparator): Participants will be maintained on 0 mg of Pioglitazone (PIO) prior to sessions assessing the abuse liability of heroin.
  Interventions: Drug: Placebo
- PIO low dose - Heroin (Experimental): Participants will be maintained on 15 mg of PIO prior to sessions assessing the abuse liability of heroin.
  Interventions: Drug: PIO
- PIO high dose - Heroin (Experimental): Participants will be maintained on 45 mg of PIO prior to sessions assessing the abuse liability of heroin.
  Interventions: Drug: PIO
- Placebo - Nicotine (Placebo Comparator): Participants will be maintained on 0 mg of PIO prior to sessions assessing the abuse liability of nicotine.
  Interventions: Drug: PIO
- PIO Low Dose - Nicotine (Experimental): Participants will be maintained on 15 mg of PIO prior to sessions assessing the abuse liability of nicotine
  Interventions: Drug: PIO
- PIO High Dose - Nicotine (Experimental): Participants will be maintained on 45 mg of PIO prior to sessions assessing the abuse liability of nicotine
  Interventions: Drug: PIO

INTERVENTIONS:
Drug: PIO — 0, 15, and 45 mg per day.
  Other Names: Actos
  Arms: PIO High Dose - Nicotine; PIO Low Dose - Nicotine; PIO high dose - Heroin; PIO low dose - Heroin; Placebo - Nicotine
Drug: Placebo — Placebo
  Other Names: Actos
  Arms: Placebo - Heroin

SUMMARY:
The goal of the proposed research is to improve the effectiveness of treatments for opioid and for nicotine dependence by testing a novel pharmacological strategy. Specifically, pioglitazone, a peroxisome proliferator-activated gamma receptor (PPARγ) agonist, will be used as an adjunct to agonist-based treatment.

DETAILED DESCRIPTION:
Although treatments for opioid and for nicotine dependence exist, these medications are not universally effective as many patients are unable to stop using or relapse rapidly, suggesting that treatment with a single agent alone is insufficient to facilitate cessation of use in many patients. Targeting additional pathways that may contribute to the maintenance of drug-taking behaviors or relapse may be a more effective strategy to treat individuals resistant to first-line approaches.

ELIGIBILITY:
Inclusion Criteria:

* 21-55 years of age
* Physically healthy
* Able to perform study procedures

Exclusion Criteria:

* Pregnancy
* Physical dependence on any other drugs besides caffeine, heroin and nicotine

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D. Comer, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented at conferences and published in a peer-reviewed journal.

REFERENCES:
- [Derived] Martinez S, Jones JD, Vadhan NP, Brandt L, Comer SD, Bisaga A. The acute and repeated effects of cigarette smoking and smoking-related cues on impulsivity. Drug Alcohol Rev. 2021 Jul;40(5):864-868. doi: 10.1111/dar.13206. Epub 2020 Nov 2. PMID 33140460

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo - Heroin: Control condition for active arms.
  Placebo: Placebo - Heroin
- Pio Low Dose - Heroin; Pio Low Dose - Nicotine: Low dose pio comparator.
  Pioglitazone: 0, 15, and 45 mg per day.
- Pio High Dose - Heroin; Pio High Dose - Nicotine: High dose pio comparator.
  Pioglitazone: 0, 15, and 45 mg per day.
- Placebo - Nicotine: Control condition for active arms.
  Pioglitazone: 0, 15, and 45 mg per day.
Period: Overall Study
Arm/Group | Placebo - Heroin | Pio Low Dose - Heroin | Pio High Dose - Heroin | Placebo - Nicotine | Pio Low Dose - Nicotine | Pio High Dose - Nicotine
Started | 19 | 4 | 18 | 15 | 9 | 17
Completed | 16 | 3 | 14 | 13 | 7 | 14
Not Completed | 3 | 1 | 4 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Heroin | Pio Low Dose - Heroin | Pio High Dose - Heroin | Placebo - Nicotine | Pio Low Dose - Nicotine | Pio High Dose - Nicotine | Total
Number analyzed (Participants) | 19 | 4 | 18 | 15 | 9 | 17 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 4 | 18 | 15 | 9 | 17 | 82
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2 | 1 | 2 | 7
  Male | 19 | 4 | 16 | 13 | 8 | 15 | 75
Region of Enrollment [Number; unit: participants]
  United States | 19 | 4 | 18 | 15 | 9 | 17 | 82

OUTCOME MEASURES:

1. Primary Outcome: Drug's Break Point
Description: Number of operant responses (mouse clicks) participants were willing to provide in order to receive the drug under investigation (heroin or nicotine). The Breakpoint is the point at which participants stopped responding for the drug, i.e., the total number of clicks they were willing to provide in order to receive the drug.
Time Frame: Following 2 weeks of Pioglitazone (PIO) maintenance.
Measure: Mean (Standard Deviation); unit: Mouse clicks
Groups:
- Pio Low Dose- Heroin: Low dose of Pio comparator
- Pio Low Dose- Nicotine: Low dose Pio comparator.
Arm/Group | Placebo - Heroin | Pio Low Dose- Heroin | Pio High Dose - Heroin | Placebo - Nicotine | Pio Low Dose- Nicotine | Pio High Dose - Nicotine
Number analyzed (Participants) | 16 | 3 | 14 | 13 | 7 | 14
Mouse clicks | 1037 (1763) | 1200 (272) | 2014 (2835) | 568 (652) | 722 (823) | 960 (1004)

2. Secondary Outcome: Measures of Subjective Drug Effects Most Commonly Indicative of Abuse Liability.
Description: Visual analog scale ratings of "Liking" reported by the participant will be the primary endpoint (0-100 mm, 0=Not at all, 100=Extremely).
Time Frame: Following 2 weeks of Pioglitazone (PIO) maintenance.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo - Heroin: Participants will be maintained on 0 mg of PIO prior to sessions assessing the abuse liability of heroin.
  Placebo: Placebo
- Pio Low Dose- Heroin: Participants will be maintained on 15 mg of PIO prior to assessing the abuse liability of heroin.
- Pio Low Dose- Nicotine: Participants will be maintained on 15 mg of PIO prior to assessing the abuse liability of nicotine.
Arm/Group | Placebo - Heroin | Pio Low Dose- Heroin | Pio High Dose - Heroin | Placebo - Nicotine | Pio Low Dose- Nicotine | Pio High Dose - Nicotine
Number analyzed (Participants) | 16 | 3 | 14 | 13 | 7 | 14
units on a scale | 24 (13) | 15 (9) | 19 (6) | 59 (9) | 68 (12) | 62.5 (10)

ADVERSE EVENTS:
Arm/Group | Placebo - Heroin | Pio Low Dose - Heroin | Pio High Dose - Heroin | Placebo - Nicotine | Pio Low Dose - Nicotine | Pio High Dose - Nicotine
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/4 | 0/18 | 0/15 | 0/9 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/4 | 0/18 | 0/15 | 0/9 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No